CLINICAL TRIAL: NCT06463158
Title: A Phase I Clinical Trial Evaluating the Impact of the Family Room App on Caregiver Well-being, Satisfaction, and Engagement in the Intensive Care Unit
Brief Title: The Impact of the Family Room App on Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 0221-24-EP
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Well-Being, Psychological; Engagement; Satisfaction, Consumer
MeSH Terms: conditions — Psychological Well-Being; Consumer Behavior

STUDY DESIGN:
Intervention Model Description: A clinical trial using a 2-stage sequential cohort design to test the impact of the Family Room on family caregiver well-being, engagement, and satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group - No Intervention (No Intervention): During the first eight months, participants will be enrolled into the control group which consists of routine care and informational practices by the intensive care unit (ICU) team.
- Intervention Group - Family Room Application (Experimental): During the last 10 months, participants will be enrolled into the intervention group where they will use the Family Room application on their personal devices.
  Interventions: Device: Family Room Application

INTERVENTIONS:
Device: Family Room Application — The Family Room application is a point of care tool that guides families on contributing to patient participant care by providing real time education, a sense of connection, emotional support, and resources that enable meaningful care giving. Importantly, family caregiver participants receive virtual training on comfort-focused care activities that can be done at the bedside, as well as a mechanism within the electronic health record (EHR) to measure and record the effectiveness of the care they provide.
  Arms: Intervention Group - Family Room Application

SUMMARY:
Engaging families in patient care during serious illness can enhance care quality, reduce social isolation, boost satisfaction, and lower healthcare costs. However, active involvement of family caregivers remains limited because there are no evidence-based tools to guide clinicians on how to include them effectively. This study will test and refine previously developed point-of-care application, Family Room, and determine its effectiveness by comparison with a control group. A series of surveys will be used to evaluate caregiver well-being, engagement and satisfaction.

DETAILED DESCRIPTION:
Engaging families in patient care during serious illness can enhance care quality, reduce social isolation, boost satisfaction, and lower healthcare costs. However, active involvement of family caregivers remains limited because there are no evidence-based tools to guide clinicians on how to include them effectively. This study will test and refine previously developed point-of-care application, Family Room, and determine its effectiveness by comparison with a control group. A series of surveys will be used to evaluate caregiver well-being, engagement and satisfaction.

The investigators will recruit participants from 5 different intensive care units (ICU) to dampen any effects experienced within a single unit. During the first 8 months of recruitment, a convenience sample of up to 50 participants (25 paired caregiver - patient dyads) will be enrolled into the control group which consists of routine care and informational practices of the ICU team. The adult family caregiver participant must be at the patient participant's bedside during ICU admission.

During the last 10 months of recruitment, up to 50 participants (25 paired caregiver - patient dyads) participants will be enrolled into the intervention group where they will use the Family Room application on their personal devices. The Family Room is a point of care tool that guides families on how to contribute to patient care by providing real time education, a sense of connection, emotional support, and resources that enable meaningful caregiving. Caregiver participants will receive virtual training on comfort-focused care activities that can be done at the bedside, as well as a mechanism within the electronic health record (EHR) to measure and record the effectiveness of the care they provide.

Data will be collected at 2 timepoints: study enrollment and within 48 hours of patient participant ICU discharge. Caregiver well-being will be measured every 48 hours while the patient participant is admitted to the ICU. Caregiver participant data will be collected through structured interviews using pre-designed questionnaires which will include items related to demographic variables, caregiver participant psychological distress, engagement, and satisfaction. Trained research assistants will conduct either face to face, virtual (via Zoom), or phone interviews depending on the caregiver participant's preference and availability. Patient participant specific data will be extracted from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Present at participant's bedside during the intensive care unit (ICU) admission
* Participant's legally authorized representative (LAR) or designated caregiver to make medical decisions on their behalf

Exclusion Criteria:

• Not legally authorized representative (LAR) or designated caregiver to make medical decisions on their behalf

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Caregiver Engagement - Practical Aspects: FAMily Engagement (FAME) Tool | At study enrollment and within 48 hours of patient participant ICU discharge
  The FAMily Engagement (FAME) questionnaire is a self-rated instrument developed to assess current family engagement. Questions address key principles of family-centered care, such as dignity and respect, information sharing, participation, and collaboration. They also address family engagement domains, including family presence, family needs, communication and education, decision making, and direct care. A five-point Likert scale (1=strongly agree, 2=agree, 3=neutral, 4=disagree, 5=strongly disagree) is used for responses, which are transformed to a 0-100 scoring system by dividing the sum of the scores by the number of questions answered. Higher scores indicate greater engagement in care and lower scores indicating lesser engagement.
Daily Activity: Family Room Application | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  The daily activity logged in the Family Room application at bedside is assessed (intervention group only).
Daily Patient Symptoms - Severity of Illness: Acute Physiology and Chronic Health Evaluation (Apache II) | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  APACHE II (Acute Physiology and Chronic Health Evaluation II) is a severity-of-disease classification system used in the ICU. An integer score is assessed by medical staff from 0 to 71 is computed based on several measurements. Higher scores correspond to more severe disease and a higher risk of death. Information is taken from the electronic health record.
Daily Patient Symptoms: Presence of Lines, Tubes and Equipment | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  A daily count of number of lines, tubes and equipment present on ICU patient participant is taken. Information is taken from the electronic health record.
Daily Patient Symptoms: Glasgow Coma Scale (GCS) | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  The Glasgow Coma Scale (GCS) is assessed by medical staff to describe the extent of impaired consciousness. Patient participants are assessed daily according to three aspects: eye-opening ("1" no response to "4" spontaneous eye opening), motor response ("1" no response to "5" oriented) and verbal response ("1" no response to "6" obeying commands). The total score ranges between 3 and 15. Higher scores indicate better responsiveness. Information is taken from the electronic health record.
Daily Patient Symptoms: Pain | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  Pain scores are assessed by medical staff daily and range from "0" (no pain) to "10" (the worst pain). Information is taken from the electronic health record.
Daily Patient Symptoms: Richmond Agitation-Sedation Scale (RASS) | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  The Richmond Agitation-Sedation Scale (RASS) is a nurse assessed 10 point scale, with -5 (unarousable) to +4 (combative). Information is taken from the electronic health record.
Daily Patient Symptoms: Confusion Assessment Method for the ICU | Daily from enrollment until patient participant ICU discharge, an average of 3 weeks
  The Confusion Assessment Method for the ICU (CAM-ICU) is a tool to assess the presence of delirium in ICU patient participant who are unable to talk. It involves a sedation assessment and a confusion assessment. The confusion assessment evaluates four features: acute onset or fluctuating course, inattention, disorganized thinking, and altered level of consciousness. A patient participant is considered to be confused if they have feature 1 plus 2 and either 3 or 4 present. The CAM-ICU score ranges from 0 to 4, with 4 being the most severe. Information is taken from the electronic health record.

SECONDARY OUTCOMES:
Caregiver Well-being: Screening Tool for Psychological Distress (STOP-D) | At study enrollment, every 48 hours while patient participant is in the ICU, and within 48 hours of patient participant ICU discharge
  This is a self-rated 5 item instrument which provides severity scores for each of the common psychosocial problem areas: depression, anxiety, stress, anger, and low social support. Scoring is "0" (not at all) to "9" (severely). The higher the score the greater the psychological distress.
Caregiver Well-being: Caregiver Self-Assessment Questionnaire | At study enrollment and within 48 hours of patient participant ICU discharge
  This is a self-rated 18-item instrument devised by the American Medical Association for physicians to assess the stress-levels of family caregivers. Caregivers are asked to respond either "Yes" or "No" to a series of statements, simple scoring system allows family caregiver themselves to score their results and to determine whether or not they are highly stressed. Points are added for each 'yes' answer for 16 questions plus a 1 to 10 score for a question of current stress levels and for a question on comparing perceived current health compared to a year ago. A higher number means more stress.
Caregiver Engagement - Psychological Experience: Caregiving Health Engagement Scale (CHE-s) | At study enrollment and within 48 hours of patient participant ICU discharge
  This is a self-rated 7 item multidimensional instrument to evaluate the impact of burden on different aspects of a caregiver's life. Caregivers respond to a series of statements, indicating their level of agreement or disagreement. The CHE is scored based on a Likert-type scale. The total score reflects the caregiver's overall engagement in healthcare. Higher scores indicate greater engagement.
Caregiver Resilience: Connor-Davidson Resilience Scale (CD-RISC2) | At study enrollment
  This is a self-rated 2 item instrument that measures resilience as it relates to ability to thrive in the face of adversity. Answers are on a 5-point scale, not true at all=0, rarely true=1, sometimes true=2, often true=3, and true nearly all of the time=4. Higher scores indicating greater perceived resilience.
Caregiver Preparedness: Preparedness for Caregiving Scale | Within 48 hours of patient participant ICU discharge
  The Preparedness for Caregiving Scale is a self-rated 10 item instrument that asks caregivers how well prepared they believe they are for multiple domains of care giving. Preparedness is defined as perceived readiness for multiple domains of the care giving role such as providing physical care, providing emotional support, setting up in-home support services, and dealing with the stress of care giving. Responses are rated on a 5-point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score the more prepared the caregiver feels for caregiving; the lower the score the less prepared the caregiver feels.

CONTACTS AND LOCATIONS:
Overall Officials: Breanna Hetland, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Nebraska Medicine, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Hetland BD, McAndrew NS, Kupzyk KA, Krutsinger DC, Pozehl BJ, Heusinkvelt JM, Camenzind CE. Family Caregiver Preferences and Contributions Related to Patient Care in the ICU. West J Nurs Res. 2022 Mar;44(3):214-226. doi: 10.1177/01939459211062954. Epub 2021 Dec 14. PMID 34904483
- [Background] Olding M, McMillan SE, Reeves S, Schmitt MH, Puntillo K, Kitto S. Patient and family involvement in adult critical and intensive care settings: a scoping review. Health Expect. 2016 Dec;19(6):1183-1202. doi: 10.1111/hex.12402. Epub 2015 Sep 7. PMID 27878937
- [Background] Kleinpell R, Heyland DK, Lipman J, Sprung CL, Levy M, Mer M, Koh Y, Davidson J, Taha A, Curtis JR; Council of the World Federation of Societies of Intensive and Critical Care Medicine. Patient and family engagement in the ICU: Report from the task force of the World Federation of Societies of Intensive and Critical Care Medicine. J Crit Care. 2018 Dec;48:251-256. doi: 10.1016/j.jcrc.2018.09.006. Epub 2018 Sep 8. PMID 30245366
- [Background] Kleinpell R, Zimmerman J, Vermoch KL, Harmon LA, Vondracek H, Hamilton R, Hanson B, Hwang DY. Promoting Family Engagement in the ICU: Experience From a National Collaborative of 63 ICUs. Crit Care Med. 2019 Dec;47(12):1692-1698. doi: 10.1097/CCM.0000000000004009. PMID 31567354
- [Background] Hetland B, Hickman R, McAndrew N, Daly B. Factors Influencing Active Family Engagement in Care Among Critical Care Nurses. AACN Adv Crit Care. 2017 Summer;28(2):160-170. doi: 10.4037/aacnacc2017118. PMID 28592476
- [Background] Hetland BD, McAndrew NS, Kupzyk KA, Krutsinger DC, Turnbull AE, Pozehl BJ, Heusinkvelt JM. Relationships among Demographic, Clinical, and Psychological Factors Associated with Family Caregiver Readiness to Participate in Intensive Care Unit Care. Ann Am Thorac Soc. 2022 Nov;19(11):1881-1891. doi: 10.1513/AnnalsATS.202106-651OC. PMID 35649201
- [Background] Hetland B, McAndrew N, Perazzo J, Hickman R. A qualitative study of factors that influence active family involvement with patient care in the ICU: Survey of critical care nurses. Intensive Crit Care Nurs. 2018 Feb;44:67-75. doi: 10.1016/j.iccn.2017.08.008. Epub 2017 Nov 21. PMID 29169879
- [Background] Tracy MF, Chlan L. Nonpharmacological interventions to manage common symptoms in patients receiving mechanical ventilation. Crit Care Nurse. 2011 Jun;31(3):19-28. doi: 10.4037/ccn2011653. PMID 21632591
- [Background] Puntillo KA, Arai S, Cohen NH, Gropper MA, Neuhaus J, Paul SM, Miaskowski C. Symptoms experienced by intensive care unit patients at high risk of dying. Crit Care Med. 2010 Nov;38(11):2155-60. doi: 10.1097/CCM.0b013e3181f267ee. PMID 20711069
- [Background] Mitchell M, Chaboyer W, Burmeister E, Foster M. Positive effects of a nursing intervention on family-centered care in adult critical care. Am J Crit Care. 2009 Nov;18(6):543-52; quiz 553. doi: 10.4037/ajcc2009226. PMID 19880956
- [Background] Mitchell ML, Kean S, Rattray JE, Hull AM, Davis C, Murfield JE, Aitken LM. A family intervention to reduce delirium in hospitalised ICU patients: A feasibility randomised controlled trial. Intensive Crit Care Nurs. 2017 Jun;40:77-84. doi: 10.1016/j.iccn.2017.01.001. Epub 2017 Feb 27. PMID 28254205
- [Background] Blom H, Gustavsson C, Sundler AJ. Participation and support in intensive care as experienced by close relatives of patients: a phenomenological study. Intensive Crit Care Nurs. 2013 Feb;29(1):1-8. doi: 10.1016/j.iccn.2012.04.002. Epub 2012 Jun 28. PMID 22748280
- [Background] Puntillo K, Arai SR, Cooper BA, Stotts NA, Nelson JE. A randomized clinical trial of an intervention to relieve thirst and dry mouth in intensive care unit patients. Intensive Care Med. 2014 Sep;40(9):1295-302. doi: 10.1007/s00134-014-3339-z. Epub 2014 Jun 4. PMID 24894026
- [Background] Yen PY, Kellye M, Lopetegui M, Saha A, Loversidge J, Chipps EM, Gallagher-Ford L, Buck J. Nurses' Time Allocation and Multitasking of Nursing Activities: A Time Motion Study. AMIA Annu Symp Proc. 2018 Dec 5;2018:1137-1146. eCollection 2018. PMID 30815156
- [Background] Choi J, Donahoe MP, Hoffman LA. Psychological and Physical Health in Family Caregivers of Intensive Care Unit Survivors: Current Knowledge and Future Research Strategies. J Korean Acad Nurs. 2016 Apr;46(2):159-67. doi: 10.4040/jkan.2016.46.2.159. PMID 27182013
- [Background] Brown SM, Rozenblum R, Aboumatar H, Fagan MB, Milic M, Lee BS, Turner K, Frosch DL. Defining patient and family engagement in the intensive care unit. Am J Respir Crit Care Med. 2015 Feb 1;191(3):358-60. doi: 10.1164/rccm.201410-1936LE. No abstract available. PMID 25635496
- [Background] Mitchell ML, Coyer F, Kean S, Stone R, Murfield J, Dwan T. Patient, family-centred care interventions within the adult ICU setting: An integrative review. Aust Crit Care. 2016 Nov;29(4):179-193. doi: 10.1016/j.aucc.2016.08.002. Epub 2016 Sep 1. PMID 27592540
- [Background] van Beusekom I, Bakhshi-Raiez F, de Keizer NF, Dongelmans DA, van der Schaaf M. Reported burden on informal caregivers of ICU survivors: a literature review. Crit Care. 2016 Jan 21;20:16. doi: 10.1186/s13054-016-1185-9. PMID 26792081
- [Background] Lindeman DA, Kim KK, Gladstone C, Apesoa-Varano EC. Technology and Caregiving: Emerging Interventions and Directions for Research. Gerontologist. 2020 Feb 14;60(Suppl 1):S41-S49. doi: 10.1093/geront/gnz178. PMID 32057082
- [Background] Adler R, Mehta R. Catalyzing technology to support family caregiving. https://www.caregivin g.org/wp-content/uploads/2020/05/Catalyzing-Technology-to-Support-FamilyCaregiving_FINAL.pdf. Updated 2014. Accessed March 31, 2022.
- [Background] Health Information and Management Systems Society. Caregiver burnout: How technology brings help and hope. https://www.himss.org/resources/caregiver-burnout-how-technologybrings-help-and-hope. Updated 2020. Accessed March 31, 2022
- [Background] Weis A, Pohlmann S, Poss-Doering R, Strauss B, Ullrich C, Hofmann H, Ose D, Winkler EC, Szecsenyi J, Wensing M. Caregivers' role in using a personal electronic health record: a qualitative study of cancer patients and caregivers in Germany. BMC Med Inform Decis Mak. 2020 Jul 13;20(1):158. doi: 10.1186/s12911-020-01172-4. PMID 32660600
- [Background] Barello S, Castiglioni C, Bonanomi A, Graffigna G. The Caregiving Health Engagement Scale (CHE-s): development and initial validation of a new questionnaire for measuring family caregiver engagement in healthcare. BMC Public Health. 2019 Nov 27;19(1):1562. doi: 10.1186/s12889-019-7743-8. PMID 31771546
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Miro. Accessed November 9, 2023. https://miro.com/
- [Background] Figma. Accessed November 9, 2023. https://www.figma.com/
- [Background] Notably. Accessed November 9, 2023. https://www.notably.ai/
- [Background] Cook TD, Campbell DT. Quasi-Experimentation: Design and analysis for field settings. Boston: Houghton Mifflin Company; 1979.
- [Background] Irmansyah I, Dharmono S, Maramis A, Minas H. Determinants of psychological morbidity in survivors of the earthquake and tsunami in Aceh and Nias. Int J Ment Health Syst. 2010 Apr 27;4(1):8. doi: 10.1186/1752-4458-4-8. PMID 20423505
- [Background] Vaishnavi S, Connor K, Davidson JR. An abbreviated version of the Connor-Davidson Resilience Scale (CD-RISC), the CD-RISC2: psychometric properties and applications in psychopharmacological trials. Psychiatry Res. 2007 Aug 30;152(2-3):293-7. doi: 10.1016/j.psychres.2007.01.006. Epub 2007 Apr 25. PMID 17459488
- [Background] Young QR, Nguyen M, Roth S, Broadberry A, Mackay MH. Single-item measures for depression and anxiety: Validation of the Screening Tool for Psychological Distress in an inpatient cardiology setting. Eur J Cardiovasc Nurs. 2015 Dec;14(6):544-51. doi: 10.1177/1474515114548649. Epub 2014 Aug 19. PMID 25139467
- [Background] Epstein-Lubow G, Gaudiano BA, Hinckley M, Salloway S, Miller IW. Evidence for the validity of the American Medical Association's caregiver self-assessment questionnaire as a screening measure for depression. J Am Geriatr Soc. 2010 Feb;58(2):387-8. doi: 10.1111/j.1532-5415.2009.02701.x. No abstract available. PMID 20370867
- [Background] Goldfarb M, Debigare S, Foster N, Soboleva N, Desrochers F, Craigie L, Burns KEA. Development of a Family Engagement Measure for the Intensive Care Unit. CJC Open. 2022 Aug 5;4(11):1006-1011. doi: 10.1016/j.cjco.2022.07.015. eCollection 2022 Nov. PMID 36444373
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] McAndrew NS, Jerofke-Owen T, Fortney CA, Costa DK, Hetland B, Guttormson J, Harding E. Systematic review of family engagement interventions in neonatal, paediatric, and adult ICUs. Nurs Crit Care. 2022 May;27(3):296-325. doi: 10.1111/nicc.12564. Epub 2020 Oct 21. PMID 33089659
- [Background] Hetland BD, Pozehl B, Kupzyk K, et al. The impact of family caregiver psychophysiological characteristics on the caregiver role in the intensive care unit. Am J Respir Crit Care Med. https://doi.org/10.1164/ajrccmconference.2019.199.1_MeetingAbstracts.A4361
- [Background] Hetland B, Bach C, Castner JP, et al. A randomized clinical trial to test a mobile application that supports family caregiver participation in patient care in the intensive care unit. Am J Respir Crit Care Med. 2023;207:A2507.
- [Background] Hetland B, Bach C, Grotts E, et al. Development of a Mobile Application to Promote Family Caregiver Engagement in the Assessment and Management of Patient Symptoms During Mechanical Ventilation in the Intensive Care Unit (ICU). Am J Respir Crit Care Med. 2021;203:A1090.
- [Background] Wilk, C. Development and Psychometric Performance of the Family Willingness for Caregiving Scale (FWCS). [Doctoral dissertation]. Kent, OH: Kent State; 2023.